CLINICAL TRIAL: NCT02540668
Title: Effect of LY3314814 on the Pharmacokinetics of Warfarin in Healthy Subjects
Brief Title: A Drug Interaction Study of Lanabecestat (LY3314814) and Warfarin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 16008; I8D-MC-AZEO (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-09-02; First posted 2015-09-04 (Estimated); Results first posted 2019-03-25 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Healthy
MeSH Terms: interventions — lanabecestat; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Warfarin (Experimental): Single oral dose of 15 mg warfarin on Day 1.
  Interventions: Drug: Warfarin
- Lanabecestat + Warfarin (Experimental): Lanabecestat administered orally once daily on Days 8 to 27, with a single oral dose of 15 mg warfarin co-administered on Day 22.
  Interventions: Drug: Lanabecestat; Drug: Warfarin

INTERVENTIONS:
Drug: Lanabecestat — Administered orally
  Other Names: LY3314814; AZD3293
  Arms: Lanabecestat + Warfarin
Drug: Warfarin — Administered orally

SUMMARY:
The purpose of this study is to look at how much warfarin gets into the blood stream and how long it takes the body to get rid of it when given both with and without lanabecestat. Another purpose is to evaluate the effectiveness of warfarin therapy to prevent blood clots when given with lanabecestat by measuring international normalized ratio (INR). INR measures the time it takes for blood to clot and compares it to an average. Information about any side effects that may occur will also be collected. The study will last about 5 weeks from the first dose to follow-up for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Male participants: will be sterile (including vasectomy) or agree to use an effective method of birth control and will not donate sperm during the study and for 3 months following the last dose of the investigational product
* Female participants: women not of childbearing potential

Exclusion Criteria:

* Have a history of or current, significant ophthalmic disease, as determined by the investigator or ophthalmologist
* Have vitiligo or any other clinically significant disorder of skin pigmentation as determined by the investigator or dermatologist
* Have a history or presence of significant bleeding disorders
* Have a history of gastrointestinal ulcers with hemorrhage
* Have a personal or family history of coagulation or bleeding disorders or reasonable suspicion of vascular malformations
* Self-reported history of increased bleeding from trauma
* Have a history of major head trauma (with loss of consciousness) within the past year or minor head trauma (without loss of consciousness) within the last 3 months prior to screening
* History of major surgery within 3 months of screening
* Planned surgery within 14 days after the last day of dosing
* International Normalized Ratio (INR)/ Prothrombin Time (PT) or activated partial thromboplastin time above the normal reference range at screening
* Abnormal Protein S antigen and/or Protein C activity as determined by the investigator
* History of deep vein thrombosis and/or pulmonary embolism

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2016-01-31 (Actual); Study Completion 2016-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Inc, Evansville, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Warfarin: Single oral dose of 15 milligram (mg) warfarin on Day 1.
- LY3314814 + Warfarin: LY3314814 administered orally once daily on Days 8 to 27, with a single oral dose of 15 mg warfarin co-administered on Day 22.
Period: Period 1 - Warfarin Single Dose
Arm/Group | Warfarin | LY3314814 + Warfarin
Started | 15 | 0
Received at Least One Dose of Study Drug | 15 | 0
Completed | 15 | 0
Not Completed | 0 | 0
Period: Period 2 - LY3314814 and Warfarin
Arm/Group | Warfarin | LY3314814 + Warfarin
Started | 0 (Warfarin was administered alone only in Period 1.) | 15 (Warfarin was co-administered with LY3314814 only in Period 2.)
Completed | 0 | 14
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who received one dose of study drug.
Groups:
- Overall: Overall study population.
Arm/Group | Overall
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 9
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Unbound S-Warfarin
Time Frame: Predose, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, and 144 hours after administration of warfarin on Days 1 and 22
Population: All participants who received at least one dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Warfarin: Single oral dose of 15 mg warfarin on Day 1. Warfarin: Administered orally
- LY3314814 + Warfarin: LY3314814 administered orally once daily on Days 8 to 27, with a single oral dose of 15 mg warfarin co-administered on Day 22. LY3314814: Administered orally Warfarin: Administered orally
Arm/Group | Warfarin | LY3314814 + Warfarin
Number analyzed (Participants) | 15 | 15
nanogram per milliliter (ng/mL) | 3.50 (12) | 3.73 (14)

2. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Curve 0-∞ (AUC) of Unbound S-Warfarin
Time Frame: Predose, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, and 144 hours after administration of warfarin on Days 1 and 22
Population: All participants who received at least one dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram * hour per milliliter(ng*h/mL)
Arm/Group | Warfarin | LY3314814 + Warfarin
Number analyzed (Participants) | 15 | 15
nanogram * hour per milliliter(ng*h/mL) | 108 (18) | 123 (19)

3. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Unbound R-Warfarin
Time Frame: Predose, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, and 144 hours after administration of warfarin on Days 1 and 22
Population: All participants who received at least one dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Warfarin | LY3314814 + Warfarin
Number analyzed (Participants) | 15 | 15
ng/mL | 4.45 (11) | 4.80 (14)

4. Secondary Outcome: Pharmacokinetics (PK): Area Under The Concentration Curve 0-∞(AUC) of Unbound R-Warfarin
Time Frame: Predose, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96,120, and 144 hours after administration of warfarin on Days 1 and 22
Population: All participants who received at least one dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Warfarin | LY3314814 + Warfarin
Number analyzed (Participants) | 15 | 15
ng*h/mL | 262 (18) | 296 (18)

5. Secondary Outcome: Pharmacodynamics (PD): Area Under the International Normalized Ratio (INR) Versus Time Curve (AUCINR) of Warfarin
Time Frame: Predose, 6, 8, 12, 24, 36, 48, 72, 96, 120, and 144 hours after administration of warfarin on Days 1 and 22
Population: All participants who received at least one dose of study drug and had evaluable pharmacodynamic INR data on Day 22 of Period 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Warfarin | LY3314814 + Warfarin
Number analyzed (Participants) | 15 | 14
ng*h/mL | 160 (9) | 158 (6)

6. Secondary Outcome: Pharmacodynamics (PD): Maximum Observed INR Response (INRmax) of Warfarin
Time Frame: Predose, 6, 8, 12, 24, 36, 48, 72, 96, 120, and 144 hours after administration of warfarin on Days 1 and 22
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Warfarin | LY3314814 + Warfarin
Number analyzed (Participants) | 15 | 14
ng/mL | 1.29 (18) | 1.26 (12)

ADVERSE EVENTS:
Groups:
- LY3314814: LY3314814 administered orally once daily on Days 8 to 27 LY3314814: Administered orally
- LY3314814 + Warfarin: Single oral dose of 15 mg warfarin co-administered on Day 22. LY3314814: Administered orally Warfarin: Administered orally
Arm/Group | Warfarin | LY3314814 | LY3314814 + Warfarin
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/15 | 1/15 | 1/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Warfarin (N=15) | LY3314814 (N=15) | LY3314814 + Warfarin (N=15)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days